CLINICAL TRIAL: NCT04159701
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 2 Crossover Study to Evaluate the Efficacy and Safety of LY3454738 in Adults With Chronic Spontaneous Urticaria Inadequately Controlled With H1-Antihistamines
Brief Title: A Study of LY3454738 in Adults With Chronic Spontaneous Urticaria
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated for lack of efficacy after an interim analysis was performed
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 17480; J1B-MC-FRCF (Other: Eli Lilly and Company); 2019-002495-13 (EudraCT Number)
Record Dates: First submitted 2019-11-08; First posted 2019-11-12 (Actual); Results first posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3454738 (Experimental): 500 milligram (mg) LY3454738 administered intravenously (IV).
  Interventions: Drug: LY3454738
- Placebo (Placebo Comparator): Placebo administered IV.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3454738 — Administered IV
  Arms: LY3454738
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
The reason for this study is to see if the study drug LY3454738 is safe and effective as treatment for participants with hives that are caused by chronic spontaneous urticaria (CSU) and that are not controlled with H1-antihistamines.

ELIGIBILITY:
Inclusion Criteria:

* Must agree to use appropriate birth control throughout the study
* Must have a diagnosis of CSU for at least 6 months
* Must have CSU symptoms for at least 8 consecutive weeks despite taking anti-histamines
* Must agree to take an anti-histamine every day during the trial
* Must be willing to enter information about symptoms in an electronic diary twice a day

Exclusion Criteria:

* Must not have a cause, other than CSU, for itching, hives, and/or angioedema (swelling beneath the skin)
* Must not have a current or recent active infection requiring antibiotics
* Must not have a history of anaphylaxis (severe, life threatening allergic reaction)
* Must not have asthma requiring medications other than short acting beta agonists (albuterol, etc.)
* Must not have received prior treatment with omalizumab, ligelizumab, or other experimental biologic for CSU

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (25):
- United States (18):
  - Kern Research, Inc, Bakersfield, California
  - First OC Dermatology, Fountain Valley, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - California Allergy and Asthma Medical Group + Research Center, Los Angeles, California
  - Allergy & Asthma Consultants, Redwood City, California
  - Florida Center for Allergy & Asthma Research Landman, Aventura, Florida
  - Florida Center for Allergy & Asthma Research Rodicio, Miami, Florida
  - Miami Dermatology and Laser Research, Miami, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - ForCare Clinical Research, Tampa, Florida
  - University of South Florida Asthma, Allergy and Immunology, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Allergy & Asthma Specialists, P.S.C., Owensboro, Kentucky
  - Johns Hopkins Asthma and Allergy Center, Baltimore, Maryland
  - Signature Allergy & Immunology, St Louis, Missouri
  - Optimed Research, LTD, Columbus, Ohio
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Northwest Research Center, Portland, Oregon
- Germany (5):
  - Medizinische Hochschule Hanover, Hanover, Lower Saxony
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz, Rhineland-Palatinate
  - Charité Campus Virchow-Klinikum, Berlin
  - Rothhaar Studien GmbH, Berlin
- Poland (2):
  - Diamond Clinic, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Evimed, Warsaw, Masovian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of LY3454738 in Adults With Chronic Spontaneous Urticaria — https://www.lillytrialguide.com/en-US/studies/hives/FRCF#?postal=

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence Group 1: (500 mg LY3454738, Placebo): Participants received 500 milligram (mg) LY3454738 intravenously (IV) every 2 weeks (Q2W) for 12 weeks followed by placebo for 12 weeks.
  Participants did not receive study drug during the follow-up period.
- Sequence Group 2: (Placebo, 500 mg LY3454738): Participants received Placebo for 12 weeks followed by 500 mg LY3454738 IV Q2W for 12 weeks.
  Participants did not receive study drug during the follow-up period.
Period: Period 1: Treatment Period
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738)
Started | 39 | 13
Received at Least One Dose of Study Drug | 39 | 13
Completed | 31 | 12
Not Completed | 8 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Study Terminated by sponsor | 4 | 1
Not completed — Withdrawal by Subject | 3 | 0
Period: Washout Period
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738)
Started | 31 | 12
Completed | 18 | 8
Not Completed | 13 | 4
Not completed — site terminated by sponsor | 0 | 1
Not completed — study terminated by sponsor | 10 | 3
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Inadvertent Enrollment | 1 | 0
Not completed — Miscellaneous | 1 | 0
Period: Period 2: Treatment Period (Crossover)
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738)
Started | 18 | 8
Completed | 18 | 5
Not Completed | 0 | 3
Not completed — Study Terminated by Sponsor | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Period: Post-treatment Follow-up
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738)
Started | 29 (All participants who received study drug could move to post-treatment follow-up.) | 9 (All participants who received study drug could move to post-treatment follow-up.)
Completed | 19 | 6
Not Completed | 10 | 3
Not completed — Study Terminated by Sponsor | 6 | 3
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Inadvertent Enrollment | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Sequence Group 1: (500 mg LY3454738, Placebo): Participants received 500 mg LY3454738 intravenously (IV) every 2 weeks (Q2W) for 12 weeks followed by placebo for 12 weeks.
- Sequence Group 2: (Placebo, 500 mg LY3454738): Participants received Placebo for 12 weeks followed by 500 mg LY3454738 IV Q2W for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738) | Total
Number analyzed (Participants) | 39 | 13 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 13 | 51
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 11 | 41
  Male | 9 | 2 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 33 | 13 | 46
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 10 | 43
  Poland | 5 | 1 | 6
  Germany | 1 | 2 | 3
Urticaria Activity Score Over 7 Days (UAS7) Score [Mean (Standard Deviation); unit: units on a scale] — The baseline UAS7 is the sum of the daily UAS over the 7 days prior to the first treatment. A higher UAS or higher UAS7 indicates greater urticaria disease activity.
  units on a scale | 26.51 (7.48) | 24.26 (5.23) | 25.95 (7.00)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Urticaria Activity Score Over 7 Days (UAS7)
Description: The UAS7 is the sum of the daily urticaria activity scores (UAS) over a 7-day period and ranges from 0 to 42. The daily UAS is the sum of the daily itch severity score (ISS) and daily number of hives score, and ranges from 0 to 6. The baseline UAS7 is the sum of the daily UAS over the 7 days prior to the first treatment. A higher UAS or higher UAS7 indicates greater urticaria disease activity.The ANCOVA model includes treatment as a factor and baseline UAS7 score in First 12-Week treatment period as covariates. Missing Week 12 scores will be imputed by carrying forward the participants' baseline scores (BOCF).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738)
Number analyzed (Participants) | 39 | 13
units on a scale | -6.38 (1.645) | -9.32 (2.864)
Statistical Analysis 1: Comparison: Sequence Group 1: (500 mg LY3454738, Placebo) vs Sequence Group 2: (Placebo, 500 mg LY3454738); Test type: Superiority; p = 0.380, Mixed Models Analysis; Mean Difference (Final Values) = 2.94, 95% CI 2-sided [-3.73 to 9.60]

2. Secondary Outcome: Mean Change From Baseline in Itch Severity Score Over 7 Days (ISS7)
Description: The ISS7 is the sum of the daily ISS over a 7-day period and ranges from 0 to 21. The daily ISS is the average of the morning and evening ISS on a 4-point scale of 0 (none), 1 (mild), 2 (moderate), and 3 (severe). The baseline ISS7 is the sum of the daily ISS over the 7 days prior to the first treatment. A higher ISS or higher ISS7 indicates more severe itching. The ANCOVA model includes treatment as a factor and baseline UAS7 score in First 12-Week treatment period as covariates. Missing Week 12 scores will be imputed by carrying forward the participants' baseline scores (BOCF).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738)
Number analyzed (Participants) | 39 | 13
units on a scale | -2.91 (0.780) | -4.21 (1.367)
Statistical Analysis 1: Comparison: Sequence Group 1: (500 mg LY3454738, Placebo) vs Sequence Group 2: (Placebo, 500 mg LY3454738); Test type: Superiority; p = 0.415, Mixed Models Analysis; Mean Difference (Final Values) = 1.30, 95% CI 2-sided [-1.89 to 4.50]

3. Secondary Outcome: Mean Change From Baseline in Hives Severity Score Over 7 Days (HSS7)
Description: The HSS7 is the sum of the daily number of hives over a 7-day period and ranges from 0 to 21. The daily number of hives score (also called HSS) is the average of the morning and evening number of hive scores on a four-point scale of 0 (none), 1 (between 1 and 6 hives, inclusive), 2 (between 7 and 12 hives, inclusive), and 3 (greater than 12 hives). The baseline weekly HSS7 is the sum of the HSS over the 7 days prior to the first treatment. A higher HSS or higher HSS7 indicates a greater number of hives. The ANCOVA model includes treatment as a factor and baseline UAS7 score in First 12-Week treatment period as covariates. Missing Week 12 scores will be imputed by carrying forward the participants' baseline scores (BOCF).
Time Frame: Baseline, Week 12
Population: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738)
Number analyzed (Participants) | 39 | 13
units on a scale | -3.45 (0.931) | -5.17 (1.631)
Statistical Analysis 1: Comparison: Sequence Group 1: (500 mg LY3454738, Placebo) vs Sequence Group 2: (Placebo, 500 mg LY3454738); Test type: Superiority; p = 0.369, Mixed Models Analysis; Mean Difference (Final Values) = 1.72, 95% CI 2-sided [-2.09 to 5.53]

4. Secondary Outcome: Percentage of Participants Achieving Urticaria Activity Score Over 7 Days (UAS7) ≤6 (Stratified by Baseline UAS7 (< 28 vs >= 28) Score)
Description: The UAS7 is the sum of the daily urticaria activity scores (UAS) over a 7-day period and ranges from 0 to 42. The daily UAS is the sum of the daily itch severity score (ISS) and daily number of hives score, and ranges from 0 to 6. The baseline UAS7 is the sum of the daily UAS over the 7 days prior to the first treatment. A higher UAS or higher UAS7 indicates greater urticaria disease activity.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had UAS7 ≤6.
Measure: Number; unit: percentage of participants
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738)
Number analyzed (Participants) | 39 | 13
percentage of participants | 15.4 | 23.1
Statistical Analysis 1: Comparison: Sequence Group 1: (500 mg LY3454738, Placebo) vs Sequence Group 2: (Placebo, 500 mg LY3454738); Test type: Superiority; p = 0.674, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted by baseline UAS7 (< 28 vs >= 28) score; Odds Ratio (OR) = 0.61, 95% CI 2-sided [0.14 to 2.70]

5. Secondary Outcome: Percentage of Participants Achieving Urticaria Activity Score Over 7 Days (UAS7) ≤6 (Stratified by Baseline UAS7 (< Median vs >= Median) Score)
Description: The UAS7 is the sum of the daily urticaria activity scores (UAS) over a 7-day period and ranges from 0 to 42.The daily UAS is the sum of the daily itch severity score (ISS) and daily number of hives score, and ranges from 0 to 6. The baseline UAS7 is the sum of the daily UAS over the 7 days prior to the first treatment. A higher UAS or higher UAS7 indicates greater urticaria disease activity.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug and had UAS7 ≤6.
Measure: Number; unit: percentage of participants
Arm/Group | Sequence Group 1: (500 mg LY3454738, Placebo) | Sequence Group 2: (Placebo, 500 mg LY3454738)
Number analyzed (Participants) | 39 | 13
percentage of participants | 15.4 | 23.1
Statistical Analysis 1: Comparison: Sequence Group 1: (500 mg LY3454738, Placebo) vs Sequence Group 2: (Placebo, 500 mg LY3454738); Test type: Superiority; p = 0.674, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel (CMH) test adjusted by baseline UAS7 (< median vs >= median) score; Odds Ratio (OR) = 0.59, 95% CI 2-sided [0.13 to 2.68]

6. Secondary Outcome: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to 336 Hours (AUC [0-336h]) of LY3454738
Description: Pharmacokinetics (PK): Area Under the Concentration Versus Time Curve From Time Zero to 336 Hours (AUC [0-336h]) of LY3454738
Time Frame: Before Infusion, after infusion, 1 hour after infusion and 2 hours after infusion on Day 1; Before Infusion on Day 8, 15, 29, 43, 57, 71, 85, 92, 99, 113, 127, 141, 155, 169 and Post-Treatment Follow-up
Population: All randomized participants who received at least one dose of LY3454738 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hour per milliliter( ug*h/mL)
Groups:
- 500 mg LY3454738: Participants received 500 mg LY3454738 intravenously (IV) every 2 weeks (Q2W) for 12 weeks.
Arm/Group | 500 mg LY3454738
Number analyzed (Participants) | 44
micrograms*hour per milliliter( ug*h/mL) | 53400 (49)

7. Secondary Outcome: PK: Maximum Concentration (Cmax) of LY3454738
Description: PK: Maximum Concentration (Cmax) of LY3454738
Time Frame: as for outcome 6
Population: All randomized participants who received at least one dose of LY3454738 and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | 500 mg LY3454738
Number analyzed (Participants) | 44
micrograms per milliliter (ug/mL) | 256 (30.8)

ADVERSE EVENTS:
Time Frame: Baseline Up To 28 Weeks
Groups:
- 500 mg LY3454738_First 12-Week Period; 500 LY3454738_Second 12-Week Crossover Period: Participants received 500 mg LY3454738 IV Q2W for 12 weeks.
- Placebo_First 12-Week Period; Placebo_Second 12-Week Crossover Period: Participants received Placebo IV Q2W for 12 weeks.
- Follow-Up Period: Participants did not receive study drug during the follow-up period.
Arm/Group | 500 mg LY3454738_First 12-Week Period | Placebo_First 12-Week Period | 500 LY3454738_Second 12-Week Crossover Period | Placebo_Second 12-Week Crossover Period | Follow-Up Period
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/13 | 0/8 | 0/18 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/13 | 0/8 | 0/18 | 0/38
Other Adverse Events (participants affected / at risk) | 4/39 | 4/13 | 1/8 | 7/18 | 2/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500 mg LY3454738_First 12-Week Period (N=39) | Placebo_First 12-Week Period (N=13) | 500 LY3454738_Second 12-Week Crossover Period (N=8) | Placebo_Second 12-Week Crossover Period (N=18) | Follow-Up Period (N=38)
Eczema eyelids (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated for lack of efficacy after an interim analysis was performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT04159701/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT04159701/SAP_001.pdf